CLINICAL TRIAL: NCT05470504
Title: Phase II Study of Growth Hormone Inhibition Using Pegvisomant In Severe Insulin Resistance
Brief Title: Study of Growth Hormone Inhibition Using Pegvisomant in Severe Insulin Resistance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000756; 000756-DK
Record Dates: First submitted 2022-07-16; First posted 2022-07-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Insulin Receptor Mutation; Partial Lipodystrophy
Keywords: Pegvisomant; Severe Insulin Resistance; Growth Hormone Inhibition; LIPOLYSIS
MeSH Terms: conditions — Lipodystrophy, Partial, Acquired; Insulin Resistance | interventions — pegvisomant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Other): open label pegvisomant
  Interventions: Drug: Pegvisomant

INTERVENTIONS:
Drug: Pegvisomant — 30 mg subcutaneously every day for 4 weeks.

SUMMARY:
Background:

Lipodystrophy (LD) syndromes are a group of rare disorders that affect how a person s body can store and use fat tissue. Many people with LDs become severely insulin resistant. Some people are insulin resistant because of a variant in the insulin receptor gene. Insulin resistance causes many health problems.

Objective:

To learn if blocking the effects of growth hormone in the body will help people with severe insulin resistance.

Eligibility:

Adults aged 18 to 65 years with either a known variant in the insulin receptor gene or with a diagnosis of partial LD.

Design:

Participants will have 2 hospital stays, about 1 month apart. Each stay will be 3 or 4 nights.

During each hospital stay, participants will have many tests. They will have a physical exam with blood tests. They will have all of their urine collected for a 24-hour period. They will have scans to measure their muscle, bone, and fat tissues. They will have tests to measure metabolism and insulin sensitivity. They may have an optional biopsy of fat tissue.

During the first hospital visit, participants will learn how to give themselves shots of a drug (pegvisomant) that blocks growth hormone. The drug is injected under the skin. Participants will continue to give themselves these shots once a day at home.

After the first hospital visit, participants will talk on the phone with members of the study team once each week. After 2 weeks they will have blood drawn for tests.

Participants will stop the shots after the second hospital visit.

DETAILED DESCRIPTION:
STUDY DESCRIPTION

The role of growth hormone (GH) in mediating pathological consequences of inadequate lipid storage will be studied in rare patient populations with high lipolysis and severe metabolic syndrome. Specifically, patients with partial lipodystrophy and pathogenic variants in the insulin receptor gene (INSR) will be studied before and after 1 month of administration of pegvisomant (a GH receptor blocker).

OBJECTIVES

Primary Objective:

Establish proof of concept that GH blockade reduces adipose tissue lipolysis in humans with severe insulin resistance.

Secondary Objectives:

Determine the effects of pegvisomant on lipolytic products and IGF-1.

ENDPOINTS

Primary Endpoint:

Adipose tissue lipolysis measured by glycerol and palmitate rates of appearance using stable isotope tracers.

Secondary Endpoints:

Free fatty acids (FFA), glycerol, IGF-1.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all the following criteria:

* Either

  * Known pathogenic variant in the insulin receptor gene, either dominant negative or recessive, OR
  * Clinical diagnosis of partial lipodystrophy based on reduction in adipose tissue outside the normal range in selected adipose depots (including, at a minimum, the gluteofemoral depot) with preservation of adipose tissue in other depots.
* Male or female, aged 18-70 years.
* Completed linear growth and puberty.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Use of niacin or other drugs that directly affect lipolysis within 8 weeks prior to enrollment.
* Patients taking anticoagulants (blood thinning medications).
* Use of non-steroidal anti-inflammatory medications (e.g., aspirin, ibuprofen) 2 weeks prior to the biopsy date (in patients who choose to undergo biopsy).
* Changes in medications for diabetes or dyslipidemia within 2 weeks prior to enrollment.
* Pregnancy or lactation.
* For females of reproductive potential: inability or unwillingness to use contraception during study participation and for an additional 1 month after the end of pegvisomant administration.
* For males of reproductive potential: inability or unwillingness to use condoms or other methods to ensure effective contraception with partner during the study and for an additional 1 month after the end of pegvisomant administration.
* Known allergic reactions pegvisomant or any of its components.
* Clinically significant liver disease, evidenced by any of the following:

  * ALT or AST >3 times the upper limit of normal at screening.
  * Current known liver disease other than steatohepatitis (e.g., autoimmune or viral hepatitis).
  * History of cirrhosis
* Triglycerides >1500 mg/dL (non-fasting) or >1000 mg/dL (fasting) at screening.
* In subjects with partial lipodystrophy only, Hemoglobin A1c >10% at screening.
* Any other medical condition or medication that, in the judgement of the investigator, will increase risk to the subject or impede the measurement of study outcomes.
* Inability of subject to understand or the unwillingness to sign a written informed consent document.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Glycerol rate of appearance (Ra) normalized to fat mass, Palmitate Ra normalized to fat mass | 1 month
  Estimate the magnitude and variability of the effect of pegvisomant, 30 mg subcutaneously once daily for 1 month, on adipose tissue lipolysis rate in subjects with pathogenic variants in the insulin receptor and partial lipodystrophy.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Result of the study will be disseminated to participants upon publication.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000756-DK.html